CLINICAL TRIAL: NCT02880553
Title: Disability, Perceived Social Support and Quality of Life in Multiple Sclerosis
Acronym: QUALVIE-SEP
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RDS_2016_11
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
The World Health Organization International Classification of Functioning, Disability and Health has shown that the environment can play a major role in patients' disability, and hence in their quality of life. This study considers social dimensions of quality of life, particularly family as well as social and professional networks.

ELIGIBILITY:
Inclusion Criteria:

* multiples sclerosis, according to McDonald's criteria

Exclusion Criteria:

* lack of French language proficiency
* severe cognitive impairment
* severe aphasia
* substance addiction
* psychiatric troubles (except for treated major depression)
* other severe neurologic or somatic disease
* pregnant or breast feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with all forms of multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
statistical association between perceived social support and quality of life | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Michèle MONTREUIL, PhD, Study Chair — Directrice du laboratoire de psychopathologie et neuropsychologie (LPN EA 2027), Université Paris 8
Locations (1):
- casa di cura de San Pellegrino, San Pellegrino, Italy